CLINICAL TRIAL: NCT03786445
Title: Analysis of In-hospital Emergency Team Calls in a German Tertiary Care University Hospital From 2013 to 2016
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Köln (Other)
Responsible Party: Sponsor
Other Study IDs: 5555-Emergency
Record Dates: First submitted 2018-12-13; First posted 2018-12-26 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Emergencies
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective analysis of 1,664 emergency forms from MET activities, ranging from January 2013 to December 2016. Every MET activation call via the emergency telephone number ("5555") and following emergency treatment was recorded by a standardized documentation form.

DETAILED DESCRIPTION:
Recent studies demonstrated that in-hospital emergencies are linked to a higher mortality in patients. In total, 1 out of 10 patients is suffering from an unexpected incident during the hospital stay. Therefore, establishing and developing medical emergency teams (MET) is getting more important in the future. Aim of the present study was an analysis of medical documentation, operational tactics and procedures taken by MET in a 4-year-period, ranging from 2013 to 2016. A retrospective analysis of 1,664 emergency forms from MET activities, ranging from January 2013 to December 2016. Every MET activation call via the emergency telephone number ("5555") and following emergency treatment was recorded by a standardized documentation form.

ELIGIBILITY:
Inclusion Criteria:

* all patients treated with emergencies

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients in the hospital
Sampling Method: Non-Probability Sample
Enrollment: 1664 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Death | 2013 to 2016
  Patients having in in-Hospital emergency.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schmitz J, Kerkhoff S, Sander D, Schulz G, Warnecke T, Hinkelbein J. [Deployment of the in-hospital emergency team in a tertiary care university hospital : Data analysis for the time period 2013-2016 in North-Rhine/Westphalia]. Anaesthesist. 2019 Jun;68(6):361-367. doi: 10.1007/s00101-019-0586-y. Epub 2019 Apr 10. German. PMID 30969357